CLINICAL TRIAL: NCT04362176
Title: Passive Immunity Trial for Our Nation (PassItOn)
Brief Title: Passive Immunity Trial for Our Nation to Treat COVID-19 in Hospitalized Adults
Acronym: PassItOn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Dolly Parton (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200738; 3UL1TR002243-04S3 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; Coronavirus; SARS-CoV-2
Keywords: COVID-19 drug treatment; convalescent plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1 to convalescent plasma versus lactated Ringer's solution with multivitamins. Randomization will be completed in permuted blocks and stratified by site, gender, and age. Participants, treating clinicians and outcomes assessors will all be blinded to study group assignment. Study personnel will not be blinded to the study group assignment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pathogen reduced SARS-CoV-2 convalescent plasma (Experimental): Transfusion of convalescent plasma will be administered by clinical or research personnel while the participant is hospitalized on Study Day 0. Plasma will be administered at a rate of 500 mL/hour and will be administered within 12 hours of randomization.
  Interventions: Biological: pathogen reduced SARS-CoV-2 convalescent plasma
- Placebo (Placebo Comparator): Participants randomized to the control group will receive 250mL of Lactate Ringers containing multivitamins intravenously on Day 1 as a placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: pathogen reduced SARS-CoV-2 convalescent plasma — Convalescent COVID-19 donor plasma is the liquid part of blood that is collected from patients who have recovered from COVID-19 infection. This plasma contains SARS-CoV-2 specific antibodies that may help fight the infection.
  Arms: pathogen reduced SARS-CoV-2 convalescent plasma
Biological: Placebo — Lactated Ringer's solution with multivitamins
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of convalescent donor plasma to treat COVID-19 in hospitalized adults in a randomized, placebo-controlled setting. The effect of convalescent plasma will be compared to placebo on clinical outcomes, measured using the COVID-19 7-point Ordinal Clinical Progression Outcomes Scale at Day 15, among adults with COVID-19 requiring hospitalization.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, participants confirmed to meet all eligibility criteria who have provided informed consent will be randomized 1:1 to convalescent plasma versus placebo. Transfusion of convalescent plasma or placebo will be administered by clinical or research personnel while the patient is hospitalized on Study Day 1. On Study Days 1-7, participants will be monitored for adverse reactions to the transfusion. Research personnel will also assess patients at Day 14 and Day 28; these assessments will be completed by phone if the participant has been discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Currently hospitalized or in an emergency department with anticipated hospitalization
3. Symptoms of acute respiratory infection, defined as one or more of the following:

   1. Cough
   2. Chills, or a fever (greater than 37.5° C or 99.5° F)
   3. Shortness of breath, operationalized as a patient having any of the following:

   i. Subjective shortness of breath reported by a patient or surrogate. ii. Tachypnea with respiratory rate of greater than 22 breaths per minute iii. Hypoxemia, defined as SpO2 less than 92% on room air, new receipt of supplemental oxygen to maintain SpO2 greater than or equal to 92%, or increased supplemental oxygen to maintain SpO2 greater than or equal to 92% for a patient on chronic oxygen therapy
4. Laboratory-confirmed SARS-CoV-2 infection within the past 14 days

Exclusion Criteria:

1. Prisoner
2. Unable to randomize within 14 days after onset of acute respiratory infection symptoms
3. Patient, legal representative, or physician not committed to full support (Exception: a patient who will receive all supportive care except for attempts at resuscitation from cardiac arrest will not be excluded.)
4. Inability to be contacted on Day 29-36 for clinical outcome assessment
5. Receipt of any SARS-CoV-2 passive immunity therapy, such as convalescent plasma, monoclonal antibodies, or pooled immunoglobulin, in the past 30 days
6. Contraindications to transfusion or history of prior reactions to transfused blood products
7. Plan for hospital discharge within 24 hours of enrollment
8. Previous enrollment in this trial
9. Previous laboratory-confirmed SARS-CoV-2 infection before the current illness
10. Enrollment in another clinical trial evaluating monoclonal antibodies, convalescent plasma, or another passive immunity therapy
11. Prior receipt of SARS-CoV-2 vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rice, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (26):
- United States (26):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - University of Colorado Denver, Aurora, Colorado
  - MedStar Health Research Institute/MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - University of Maryland, Baltimore (University of Maryland Medical Center), Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellelsey Hospital, Newton, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University at Buffalo/Buffalo General Medical Center, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - Cleveland Clinic Ohio, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center and James Cancer Hospital, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Utah Valley Hospital, Provo, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Rio C, Malani PN. COVID-19-New Insights on a Rapidly Changing Epidemic. JAMA. 2020 Apr 14;323(14):1339-1340. doi: 10.1001/jama.2020.3072. No abstract available. PMID 32108857
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Perlman S. Another Decade, Another Coronavirus. N Engl J Med. 2020 Feb 20;382(8):760-762. doi: 10.1056/NEJMe2001126. Epub 2020 Jan 24. No abstract available. PMID 31978944
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Cui J, Li F, Shi ZL. Origin and evolution of pathogenic coronaviruses. Nat Rev Microbiol. 2019 Mar;17(3):181-192. doi: 10.1038/s41579-018-0118-9. PMID 30531947
- [Background] Cheng PK, Wong DA, Tong LK, Ip SM, Lo AC, Lau CS, Yeung EY, Lim WW. Viral shedding patterns of coronavirus in patients with probable severe acute respiratory syndrome. Lancet. 2004 May 22;363(9422):1699-700. doi: 10.1016/S0140-6736(04)16255-7. PMID 15158632
- [Background] Hui DS, Azhar EI, Kim YJ, Memish ZA, Oh MD, Zumla A. Middle East respiratory syndrome coronavirus: risk factors and determinants of primary, household, and nosocomial transmission. Lancet Infect Dis. 2018 Aug;18(8):e217-e227. doi: 10.1016/S1473-3099(18)30127-0. Epub 2018 Apr 18. PMID 29680581
- [Background] Wang Y, Liu Y, Liu L, Wang X, Luo N, Li L. Clinical Outcomes in 55 Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Who Were Asymptomatic at Hospital Admission in Shenzhen, China. J Infect Dis. 2020 May 11;221(11):1770-1774. doi: 10.1093/infdis/jiaa119. PMID 32179910
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Wilson N, Kvalsvig A, Barnard LT, Baker MG. Case-Fatality Risk Estimates for COVID-19 Calculated by Using a Lag Time for Fatality. Emerg Infect Dis. 2020 Jun;26(6):1339-1441. doi: 10.3201/eid2606.200320. Epub 2020 Jun 17. PMID 32168463
- [Background] Niewiesk S. Maternal antibodies: clinical significance, mechanism of interference with immune responses, and possible vaccination strategies. Front Immunol. 2014 Sep 16;5:446. doi: 10.3389/fimmu.2014.00446. eCollection 2014. PMID 25278941
- [Background] Casadevall A. Passive antibody therapies: progress and continuing challenges. Clin Immunol. 1999 Oct;93(1):5-15. doi: 10.1006/clim.1999.4768. PMID 10497006
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Zhou B, Zhong N, Guan Y. Treatment with convalescent plasma for influenza A (H5N1) infection. N Engl J Med. 2007 Oct 4;357(14):1450-1. doi: 10.1056/NEJMc070359. No abstract available. PMID 17914053
- [Background] Wu XX, Gao HN, Wu HB, Peng XM, Ou HL, Li LJ. Successful treatment of avian-origin influenza A (H7N9) infection using convalescent plasma. Int J Infect Dis. 2015 Dec;41:3-5. doi: 10.1016/j.ijid.2015.10.009. Epub 2015 Oct 23. PMID 26482389
- [Background] Kraft CS, Hewlett AL, Koepsell S, Winkler AM, Kratochvil CJ, Larson L, Varkey JB, Mehta AK, Lyon GM 3rd, Friedman-Moraco RJ, Marconi VC, Hill CE, Sullivan JN, Johnson DW, Lisco SJ, Mulligan MJ, Uyeki TM, McElroy AK, Sealy T, Campbell S, Spiropoulou C, Stroher U, Crozier I, Sacra R, Connor MJ Jr, Sueblinvong V, Franch HA, Smith PW, Ribner BS; Nebraska Biocontainment Unit and the Emory Serious Communicable Diseases Unit. The Use of TKM-100802 and Convalescent Plasma in 2 Patients With Ebola Virus Disease in the United States. Clin Infect Dis. 2015 Aug 15;61(4):496-502. doi: 10.1093/cid/civ334. Epub 2015 Apr 22. PMID 25904375
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Cao J, Hu X, Cheng W, Yu L, Tu WJ, Liu Q. Clinical features and short-term outcomes of 18 patients with corona virus disease 2019 in intensive care unit. Intensive Care Med. 2020 May;46(5):851-853. doi: 10.1007/s00134-020-05987-7. Epub 2020 Mar 2. No abstract available. PMID 32123993
- [Background] Baden LR, Rubin EJ. Covid-19 - The Search for Effective Therapy. N Engl J Med. 2020 May 7;382(19):1851-1852. doi: 10.1056/NEJMe2005477. Epub 2020 Mar 18. No abstract available. PMID 32187463
- [Background] Xiao AT, Gao C, Zhang S. Profile of specific antibodies to SARS-CoV-2: The first report. J Infect. 2020 Jul;81(1):147-178. doi: 10.1016/j.jinf.2020.03.012. Epub 2020 Mar 21. No abstract available. PMID 32209385
- [Background] Haveri A, Smura T, Kuivanen S, Osterlund P, Hepojoki J, Ikonen N, Pitkapaasi M, Blomqvist S, Ronkko E, Kantele A, Strandin T, Kallio-Kokko H, Mannonen L, Lappalainen M, Broas M, Jiang M, Siira L, Salminen M, Puumalainen T, Sane J, Melin M, Vapalahti O, Savolainen-Kopra C. Serological and molecular findings during SARS-CoV-2 infection: the first case study in Finland, January to February 2020. Euro Surveill. 2020 Mar;25(11):2000266. doi: 10.2807/1560-7917.ES.2020.25.11.2000266. PMID 32209163
- [Background] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- [Background] Okba NMA, Muller MA, Li W, Wang C, GeurtsvanKessel CH, Corman VM, Lamers MM, Sikkema RS, de Bruin E, Chandler FD, Yazdanpanah Y, Le Hingrat Q, Descamps D, Houhou-Fidouh N, Reusken CBEM, Bosch BJ, Drosten C, Koopmans MPG, Haagmans BL. Severe Acute Respiratory Syndrome Coronavirus 2-Specific Antibody Responses in Coronavirus Disease Patients. Emerg Infect Dis. 2020 Jul;26(7):1478-1488. doi: 10.3201/eid2607.200841. Epub 2020 Jun 21. PMID 32267220
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wang Y, Fan G, Salam A, Horby P, Hayden FG, Chen C, Pan J, Zheng J, Lu B, Guo L, Wang C, Cao B. Comparative Effectiveness of Combined Favipiravir and Oseltamivir Therapy Versus Oseltamivir Monotherapy in Critically Ill Patients With Influenza Virus Infection. J Infect Dis. 2020 Apr 27;221(10):1688-1698. doi: 10.1093/infdis/jiz656. PMID 31822885
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Kidney Disease Improving Global Outcomes. KDIGO clinical practice guideline for acute kidney injury. Kidney Int. 2012;2: Suppl:1-138.
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Ginde AA, Brower RG, Caterino JM, Finck L, Banner-Goodspeed VM, Grissom CK, Hayden D, Hough CL, Hyzy RC, Khan A, Levitt JE, Park PK, Ringwood N, Rivers EP, Self WH, Shapiro NI, Thompson BT, Yealy DM, Talmor D. Early High-Dose Vitamin D3 for Critically Ill, Vitamin D-Deficient Patients. N Engl J Med. 2019 Dec 26;381(26):2529-2540. doi: 10.1056/NEJMoa1911124. Epub 2019 Dec 11. PMID 31826336
- [Background] Whitehead J. Sample size calculations for ordered categorical data. Stat Med. 1993 Dec 30;12(24):2257-71. doi: 10.1002/sim.4780122404. PMID 8134732
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] National Bioethics Advisory Commitee (NBAC). Research Involving Persons with Mental Disorders That May Affect Decisionmaking Capacity. U.S. Government Printing Office; 1998.
- [Background] Dresser R. Research Involving Persons with Mental Disabilities: A Review of Policy Issues and Proposals. Rockville: U.S. Government Printing Office; 1998:5-28.
- [Background] Cognitively impaired subjects. American College of Physicians. Ann Intern Med. 1989 Nov 15;111(10):843-8. No abstract available. PMID 2683918
- [Derived] Self WH, Wheeler AP, Stewart TG, Schrager H, Mallada J, Thomas CB, Cataldo VD, O'Neal HR Jr, Shapiro NI, Higgins C, Ginde AA, Chauhan L, Johnson NJ, Henning DJ, Jaiswal SJ, Mammen MJ, Harris ES, Pannu SR, Laguio-Vila M, El Atrouni W, de Wit M, Hoda D, Cohn CS, McWilliams C, Shanholtz C, Jones AE, Raval JS, Mucha S, Ipe TS, Qiao X, Schrantz SJ, Shenoy A, Fremont RD, Brady EJ, Carnahan RH, Chappell JD, Crowe JE Jr, Denison MR, Gilchuk P, Stevens LJ, Sutton RE, Thomsen I, Yoder SM, Bistran-Hall AJ, Casey JD, Lindsell CJ, Wang L, Pulley JM, Rhoads JP, Bernard GR, Rice TW; Passive Immunity Trial for Our Nation (PassITON) Investigators. Neutralizing COVID-19 Convalescent Plasma in Adults Hospitalized With COVID-19: A Blinded, Randomized, Placebo-Controlled Trial. Chest. 2022 Nov;162(5):982-994. doi: 10.1016/j.chest.2022.06.029. Epub 2022 Jul 1. PMID 35780813
- [Derived] Self WH, Stewart TG, Wheeler AP, El Atrouni W, Bistran-Hall AJ, Casey JD, Cataldo VD, Chappell JD, Cohn CS, Collins JB, Denison MR, de Wit M, Dixon SL, Duggal A, Edwards TL, Fontaine MJ, Ginde AA, Harkins MS, Harrington T, Harris ES, Hoda D, Ipe TS, Jaiswal SJ, Johnson NJ, Jones AE, Laguio-Vila M, Lindsell CJ, Mallada J, Mammen MJ, Metcalf RA, Middleton EA, Mucha S, O'Neal HR Jr, Pannu SR, Pulley JM, Qiao X, Raval JS, Rhoads JP, Schrager H, Shanholtz C, Shapiro NI, Schrantz SJ, Thomsen I, Vermillion KK, Bernard GR, Rice TW; Passive Immunity Trial for Our Nation (PassITON) Investigators. Passive Immunity Trial for Our Nation (PassITON): study protocol for a randomized placebo-control clinical trial evaluating COVID-19 convalescent plasma in hospitalized adults. Trials. 2021 Mar 20;22(1):221. doi: 10.1186/s13063-021-05171-2. PMID 33743799
- [Derived] Self WH, Stewart TG, Wheeler AP, El Atrouni W, Bistran-Hall AJ, Casey JD, Cataldo VD, Chappell JD, Cohn CS, Collins JB, Denison MR, de Wit M, Dixon SL, Duggal A, Edwards TL, Fontaine MJ, Ginde AA, Harkins MS, Harrington T, Harris ES, Hoda D, Ipe TS, Jaiswal SJ, Johnson NJ, Jones AE, Laguio-Vila M, Lindsell CJ, Mallada J, Mammen MJ, Metcalf RA, Middleton EA, Mucha S, O'Neal HR, Pannu SR, Pulley JM, Qiao X, Raval JS, Rhoads JP, Schrager H, Shanholtz C, Shapiro NI, Schrantz SJ, Thomsen I, Vermillion KK, Bernard GR, Rice TW. Passive Immunity Trial for Our Nation (PassITON): study protocol for a randomized placebo-control clinical trial evaluating COVID-19 convalescent plasma in hospitalized adults. Res Sq [Preprint]. 2021 Mar 2:rs.3.rs-227796. doi: 10.21203/rs.3.rs-227796/v1. PMID 33688640
- See also: Discovery of a novel coronavirus associated with the recent pneumonia outbreak in humans and its potential bat origin — https://www-biorxiv-org.proxy.library.vanderbilt.edu/content/10.1101/2020.01.22.914952v2
- See also: China puts 245 COVID-19 patients on convalescent plasma therapy - Xinhua — http://www.xinhuanet.com/english/2020-02/28/c_138828177.htm
- See also: WHO | Coronavirus disease (COVID-2019) R&D — https://www.who.int/blueprint/priority-diseases/key-action/novel-coronavirus/en/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Started | 495 | 479
Completed | 482 | 465
Not Completed | 13 | 14
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawn (Participant/PI withdrew consent) | 8 | 6

BASELINE CHARACTERISTICS:
Population: The 14 patients not included in the analysis all withdrew their consent following randomization which removes them from the primary analytical population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo | Total
Number analyzed (Participants) | 487 | 473 | 960
Age, Categorical [Count of Participants; unit: Participants] — Population: Final analysis only included 960 participants. The 14 patients not included in the analysis all withdrew their consent following randomization which removes them from the primary analytical population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 296 | 301 | 597
    >=65 years | 191 | 172 | 363
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 204 | 410
  Male | 281 | 269 | 550
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The 14 patients not included in the analysis all withdrew their consent following randomization which removes them from the primary analytical population.
  Participants
    Hispanic or Latino | 72 | 71 | 143
    Not Hispanic or Latino | 406 | 396 | 802
    Unknown or Not Reported | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The 14 patients not included in the analysis all withdrew their consent following randomization which removes them from the primary analytical population.
  Participants
    American Indian or Alaska Native | 6 | 5 | 11
    Asian | 14 | 11 | 25
    Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
    Black or African American | 104 | 80 | 184
    White | 272 | 285 | 557
    More than one race | 8 | 11 | 19
    Unknown or Not Reported | 81 | 77 | 158
Region of Enrollment [Number; unit: participants] — Population: The 14 patients not included in the analysis all withdrew their consent following randomization which removes them from the primary analytical population.
  participants
    United States | 487 | 473 | 960

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 7-point Ordinal Clinical Progression Outcomes Scale Score
Description: Outcome measured clinical status of the participant defined by the Covid-19 7-point Ordinal Clinical Progression Outcomes Scale: This scale reflects a range from baseline to death as follows:
  1. Not hospitalized with resumption of normal activities.
  2. Not hospitalized, but unable to resume normal activities.
  3. Hospitalized, not on supplemental oxygen.
  4. Hospitalized, on supplemental oxygen.
  5. Hospitalized, on nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both
  6. Hospitalized, on ECMO, invasive mechanical ventilation, or both.
  7. Death
Time Frame: Study Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants
  1: not hospitalized with resumption of normal pre-illness activities | 150 | 144
  2: not hospitalized but unable to resume normal pre-illness activities | 157 | 167
  3: hospitalized and not on supplemental oxygen | 16 | 11
  4: hospitalized and on standard flow oxygen | 42 | 39
  5: hospitalized and on nasal high flow oxygen therapy or non-invasive ventilation | 16 | 15
  6: hospitalized and on invasive mechanical ventilation or ECMO | 43 | 49
  7: death | 63 | 48

2. Secondary Outcome: All-location, All-cause 14-day Mortality
Description: All-location, all-cause 14-day mortality; mortality was assessed via EHR review, phone call, social media review
Time Frame: Baseline to Study Day 14
Population: The participant flow table, lists the 947 that are not lost to follow-up. This matches the N for day 14 and day 28 mortality. While the primary endpoint can be calculated from the "not withdrawn" population, the mortality endpoints come from the "not lost-to-follow-up" population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 482 | 465
Participants | 63 | 48

3. Secondary Outcome: All-location, All-cause 28-day Mortality
Description: All-location, all-cause 28-day mortality
Time Frame: Baseline to Study Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 482 | 465
Participants | 89 | 80

4. Secondary Outcome: Survival Through 28 Days
Description: Number of participants survived through Day 28
Time Frame: Baseline to Day 28 (assessed on Study Day 29)
Population: The participant flow table, lists the 947 that are not lost to follow-up. Analysis includes 482 in the Convalescent Plasma arm and 465 in the Placebo arm. This matches the N for day 14 and day 28 mortality. While the primary endpoint can be calculated from the "not withdrawn" population, the mortality endpoints come from the "not lost-to-follow-up" population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 482 | 465
Participants | 393 | 385

5. Secondary Outcome: COVID-19 7-point Ordinal Clinical Progression Outcomes Scale on Study Day 3
Description: as for outcome 1
Time Frame: Baseline to Study Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants
  1: not hospitalized with resumption of normal pre-illness activities | 1 | 6
  2: not hospitalized but unable to resume normal pre-illness activities | 49 | 54
  3: hospitalized and not on supplemental oxygen | 42 | 49
  4: hospitalized and on standard flow oxygen | 201 | 184
  5: hospitalized and on nasal high flow oxygen therapy or non-invasive ventilation | 110 | 113
  6: hospitalized and on invasive mechanical ventilation or ECMO | 74 | 63
  7: death | 10 | 4

6. Secondary Outcome: COVID-19 7-point Ordinal Clinical Progression Outcomes Scale on Study Day 8
Description: as for outcome 1
Time Frame: Study Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants
  1: not hospitalized with resumption of normal pre-illness activities | 95 | 110
  2: not hospitalized but unable to resume normal pre-illness activities | 130 | 125
  3: hospitalized and not on supplemental oxygen | 31 | 16
  4: hospitalized and on standard flow oxygen | 77 | 78
  5: hospitalized and on nasal high flow oxygen therapy or non-invasive ventilation | 58 | 60
  6: hospitalized and on invasive mechanical ventilation or ECMO | 64 | 62
  7: death | 32 | 22

7. Secondary Outcome: COVID-19 7-point Ordinal Clinical Progression Outcomes Scale on Study Day 29
Description: as for outcome 1
Time Frame: Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants
  1: not hospitalized with resumption of normal pre-illness activities | 183 | 204
  2: not hospitalized but unable to resume normal pre-illness activities | 168 | 144
  3: hospitalized and not on supplemental oxygen | 7 | 7
  4: hospitalized and on standard flow oxygen | 11 | 14
  5: hospitalized and on nasal high flow oxygen therapy or non-invasive ventilation | 5 | 4
  6: hospitalized and on invasive mechanical ventilation or ECMO | 24 | 20
  7: death | 89 | 80

8. Secondary Outcome: Oxygen-free Days Through Day 28
Description: Number of days without use of oxygen
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Day | 21 [0 to 25] | 21 [0 to 25]

9. Secondary Outcome: Ventilator-free Days Through Day 28
Description: Number of days without use of a ventilator
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Day | 28 [18 to 28] | 28 [22 to 28]

10. Secondary Outcome: Vasopressor-free Days Through Day 28
Description: Number of days without use of vasopressors
Time Frame: Baseline to Day 28
Measure: Mean (Inter-Quartile Range); unit: Day
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Day | 28 [27 to 28] | 28 [26 to 28]

11. Secondary Outcome: ICU-free Days Through Day 28
Description: Number of days outside of ICU
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Day | 28 [2 to 28] | 28 [13 to 28]

12. Secondary Outcome: Hospital-free Days Through Day 28
Description: Number of days outside of the hospital
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Day | 20 [0 to 24] | 21 [0 to 24]

13. Other Pre Specified Outcome: Acute Kidney Injury
Description: Number of participants with Acute kidney injury
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 2 | 0

14. Other Pre Specified Outcome: Renal Replacement Therapy
Description: Number of participants requiring renal replacement therapy
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 20 | 15

15. Other Pre Specified Outcome: Documented Venous Thromboembolic Disease (DVT or PE)
Description: Number of participants with documented venous thromboembolic disease (DVT or PE)
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 101 | 109

16. Other Pre Specified Outcome: Documented Cardiovascular Event (Myocardial Infarction or Ischemic Stroke)
Description: Number of Participants with myocardial infarction or ischemic stroke
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 22 | 18

17. Other Pre Specified Outcome: Transfusion Reaction
Description: Number of participants with transfusion reaction (fever/rash)
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 6 | 0

18. Other Pre Specified Outcome: Transfusion Related Acute Lung Injury (TRALI)
Description: Number of participants with transfusion related acute lung injury (TRALI)
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 0 | 0

19. Other Pre Specified Outcome: Transfusion Associated Circulatory Overload (TACO)
Description: Number of participants with transfusion associated circulatory overload (TACO)
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 1 | 0

20. Other Pre Specified Outcome: Transfusion Related Infection
Description: Number of participants with transfusion related infection
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
Number analyzed (Participants) | 487 | 473
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline - Day 90
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion
Arm/Group | Pathogen Reduced SARS-CoV-2 Convalescent Plasma | Placebo
All-Cause Mortality (participants affected / at risk) | 89/495 | 80/479
Serious Adverse Events (participants affected / at risk) | 21/495 | 16/479
Other Adverse Events (participants affected / at risk) | 27/495 | 19/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pathogen Reduced SARS-CoV-2 Convalescent Plasma (N=495) | Placebo (N=479)
acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
cardiac disorder, other, pneumopericardium (Cardiac disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Guillain-Barre Syndrome Grade 3 (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Peritoneal Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Cardiac disorders) | 0 (0) | 1 (1)
Worsening respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pathogen Reduced SARS-CoV-2 Convalescent Plasma (N=495) | Placebo (N=479)
Abdominal pain (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increase (Investigations) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blurry Vision (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders-Other, irregular heartbeat (Cardiac disorders) | 0 (0) | 1 (1)
cardiac disorders - other (volume overload) (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 3 (3) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
decompensated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 2 (2)
Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
left hand tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
nausea (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pleuritic Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sore throat (General disorders) | 0 (0) | 1 (1)
subcutaneous emphysema tracks (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
worsening hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
worsening of acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT04362176/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT04362176/SAP_002.pdf
  • Informed Consent Form (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT04362176/ICF_000.pdf